CLINICAL TRIAL: NCT02062333
Title: The Effects of the Drugs Used in Hypotensive Anaesthesia on Cochlea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Recep Aksu, associate professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/425
Record Dates: First submitted 2014-02-06; First posted 2014-02-13 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Anesthesia; Adverse Effect; Reflex, Abnormal; Tinnitus, Spontaneous Oto-Acoustic Emission
Keywords: dexmedetomidine; esmolol; stapes reflex
MeSH Terms: conditions — Reflex, Abnormal; Tinnitus | interventions — Dexmedetomidine; esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Active Comparator): 0,4-0,8 µg./kg./h dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- esmolol (Active Comparator): 100- 300 µg./kg./min esmolol
  Interventions: Drug: esmolol

INTERVENTIONS:
Drug: Dexmedetomidine — 1 mcg/kg dexmedetomidine is applied bolus and 0.2 mcg/kg/h dexmedetomidine is applied iv infusion
  Other Names: precedex
  Arms: dexmedetomidine
Drug: esmolol — 500 mcg/kg brevibloc is applied bolus and 100 mcg/kg/h iv infusion
  Other Names: breviblock
  Arms: esmolol

SUMMARY:
The aim of this study is to find the Effects of Anesthetics Used in Hypotensive Anesthesia on Stapes Reflex and Distortion Product Auto Acoustic Emission.

DETAILED DESCRIPTION:
This study was aimed at evaluating the effects of dexmedetomidine and esmolol on stapes reflex and distortion product auto acoustic emission. the stapes reflex and auto acoustic emission are of considerable diagnostic significances in otolaryngology this are objective methods for the assessment of auditory function.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 age
* American Society of Anaesthesiologists physical status classification (ASA)1-2
* tympanoplasty surgery
* patients with normal stapes reflexes

Exclusion Criteria:

* hypertension
* drug allergy
* cardiac problems
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
distortion product auto acoustic emission | postoperative 1 day
  distortion product measurements will be performed in 1001, 1501, 2002, 3003, 4004, 6006, 7996 Hz frequencies and change from baseline in distortion product measurements at postoperative 1 day

SECONDARY OUTCOMES:
stapes reflex | postoperative 1 day
  stapes muscle reflex measurements will be performed by electrical impedance. data will be taken as graphics. ıf there is an amplitude on graphic the data will be assumed as stapes reflex positive.Change from Baseline in stapes muscle reflex at postoperative 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Gunhan Gokahmetoglu, M.D, Principal Investigator — M.D
Locations (1):
- Kayseri Education and Research Hospital, Kayseri, Turkey (Türkiye)